CLINICAL TRIAL: NCT03413748
Title: Comparative Study Between Intraabdominal Irrigation and Non Irrigation During Elective Cesarean Section
Brief Title: Peritoneal Irrigation at Elective Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 23
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Postoperative Recovery
MeSH Terms: interventions — Peritoneal Lavage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peritoneal irrigation (Active Comparator): Irrigation with 500 - 1000 ml of warm normal saline will be done after closure of visceral peritoneum
  Interventions: Procedure: Elective Cesarean Section; Other: Peritoneal irrigation
- Non peritoneal irrigation (Active Comparator): No Irrigation with 500 - 1000 ml of warm normal saline will be done after closure of visceral peritoneum
  Interventions: Procedure: Elective Cesarean Section

INTERVENTIONS:
Procedure: Elective Cesarean Section — lower segment cesarean section
  Other Names: CS
Other: Peritoneal irrigation — Irrigation of peritoneal cavity with 500 - 1000 ml of warm normal saline
  Arms: Peritoneal irrigation

SUMMARY:
All participants will be randomized at elective cesarean section to either irrigation with 500 to 1000 ml of warm normal saline after closure of visceral peritoneum or non irrigation

DETAILED DESCRIPTION:
All participants will be randomized at elective cesarean section to either irrigation with 500 to 1000 ml of warm normal saline after closure of visceral peritoneum or non irrigation during the procedure of elective lower segment cesarean section

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Gestational age 36 - 40 weeks
* Elective Cesarean section
* Under spinal anaesthesia

Exclusion Criteria:

* Chronic diseases as Diabetes and hypertension
* Intestinal diseases as Crohn's disease
* Psychological and neurological conditions affecting pain sensation
* women with ferbrile morbidity before the operation
* The need for general anesthesia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Intestinal recovery | 24 hours after operation
  Auscultation of intestinal sounds

SECONDARY OUTCOMES:
Temperature | every hour for 16 hours after the operation
  measuring the oral temperature by thermometer
postoperative pain | 24 hours after surgery
  Pain score felt by the patient using Visual analogue score

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No